CLINICAL TRIAL: NCT05864248
Title: Feasibility Study SA of the Supira System for HRPCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Supira Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-10002
Record Dates: First submitted 2023-04-26; First posted 2023-05-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Heart Diseases; Coronary Artery Disease (CAD); Heart Failure
Keywords: High-risk percutaneous coronary intervention; Peripheral ventricular assist device; Supira System
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HRPCI patients (Experimental): Patients undergoing non-emergent, high-risk percutaneous coronary interventions.
  Interventions: Device: Supira System

INTERVENTIONS:
Device: Supira System — The Supira System is a temporary (≤ 4 hours) ventricular support device indicated for use during elective or urgent high-risk percutaneous coronary interventions (HRPCI) performed in hemodynamically stable patients with severe coronary artery disease when a heart team has determined HRPCI is the appropriate therapeutic option.

SUMMARY:
The objective is to assess the feasibility and safety of the Supira System in providing temporary cardiovascular hemodynamic support in patients undergoing high-risk percutaneous interventions (HRPCI).

DETAILED DESCRIPTION:
The Feasibility Study SA is a prospective, single-arm, interventional multi-center study enrolling up to 100 treated subjects.

The Supira Catheter is a single-use percutaneous expandable blood pump designed to unload the left ventricle by actively transporting blood from the left ventricle into the aorta.

The Supira System is a temporary (≤ 4 hours) ventricular support device indicated for use during elective or urgent high-risk percutaneous coronary interventions (HRPCI) performed in hemodynamically stable patients with severe coronary artery disease when a heart team has determined HRPCI is the appropriate therapeutic option

ELIGIBILITY:
To be eligible, subjects must meet ALL of the following inclusion criteria:

1. Age ≥ 18 and ≤ 90 years
2. Will undergo elective or urgent HRPCI, where hemodynamic support is needed, as determined by the institutional Heart Team
3. Signed the informed consent

To be eligible, subjects must NOT meet ANY of the following exclusion criteria:

1. Cardiogenic shock or acutely decompensated pre-existing chronic heart failure. Cardiogenic shock is defined as: systemic hypotension (systolic BP < 90 mmHg or the need for inotropes/pressors to maintain a systolic BP > 90 mmHg) plus one of the following: any requirement for inotropes/pressors prior to arrival at the catheterization laboratory, clinical evidence of end-organ hypoperfusion or use of intra-aortic balloon pump (IABP), or any other circulatory support device.
2. Stroke within 6 months of the index procedure, or any prior stroke with permanent neurologic deficit
3. Evidence of left ventricular thrombus
4. Moderate or greater aortic valvular disease or regurgitation (≥ 2+ on a 4-grade scale as assessed on transthoracic echo cardiogram (TTE)
5. Moderate or greater aortic stenosis (gradient >20 mmHg or valve area < 1.5 cm^2 as assessed on TTE)
6. Previous aortic valve replacement or reconstruction
7. Ascending or descending aortic dissection or aortic aneurysm > 4.5 cm
8. Aortic and iliofemoral anatomical conditions that preclude safe delivery and placement of the device
9. Presence of decompensated liver disease; severe liver dysfunction (Child class C)
10. Patients requiring renal replacement therapy with dialysis
11. Infection of the proposed procedural access site or systemic active infection requiring ongoing antibiotic therapy
12. Current or history of heparin-induced thrombocytopenia (HIT)
13. Known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or has known hypersensitivity to heparin, aspirin, ADP receptor inhibitors, or nitinol
14. Known or suspected coagulopathy or abnormal coagulation parameters (defined as platelet count ≤ 100,000/mm³ or spontaneous INR ≥ 1.5 or known fibrinogen ≤ 1.5 g/L)
15. Any condition or scheduled surgery that will require discontinuation of antiplatelet and/or anticoagulant therapy within 90 days of the index procedure
16. Planned coronary intervention within 30 days post index procedure
17. Breastfeeding or pregnant
18. Currently participating in active follow-up phase of another clinical study of an investigational drug or device
19. Active COVID-related infection or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
20. Subject has other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to provide written informed consent and/or to comply with study procedures
21. Considered to be part of a vulnerable population (defined as individuals with mental disability, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent; vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Endpoint: Successful initiation and maintenance of hemodynamic support without sustained hypotension throughout the index procedure. | From device delivery through device removal (up to 4 hours).
  Sustained hypotension is defined as sustained mean arterial pressure (MAP) < 60mmHg requiring (1) more than one administration of inotropes/vasopressors within 5 minutes, OR (2) continuous infusion of inotropic/pressor medications, OR 3) alternative mechanical circulatory support, to restore hemodynamics.
Primary Safety Endpoint: Rate of composite major device-related adverse events (MDRAEs), from device delivery through device removal. | From device delivery through device removal (up to 4 hours).
  MDRAEs related to the device.

SECONDARY OUTCOMES:
Rate of Technical Success. | From device delivery through device removal (up to 4 hours).
  Completion of the entire Supira System procedure, including delivery, operation without device malfunction, and successful retrieval of the catheter.
Rate of Procedural Success | From device delivery through device removal (up to 4 hours).
  Rate of technical success without procedural serious adverse events (SAEs).
Rate of composite MDRAEs from device removal through hospital discharge or 72 hours post-procedure, whichever comes first. | From device removal through hospital discharge or 72 hours post-procedure, whichever occurs first.
  MDRAEs related to the study device.
Rate of composite MDRAE from hospital discharge or 72 hours post-procedure (whichever occurs first) through 30 days post device removal. | From hospital discharge or 72 hours post-procedure (whichever occurs first)
  Major adverse events related to the study device.
Rate of composite MDRAE from 30 days to 90 days post device removal (for subjects enrolled and treated after the first 30 subjects). | From 30 days to 90 days post device removal.
  Major adverse events related to the device.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto Dante Pazzanese De Cardiologia (Dante), São Paulo
  - 'Instituto Do Coração de São Paulo (InCor)', São Paulo

IPD SHARING:
Plan to Share IPD: No